CLINICAL TRIAL: NCT05478811
Title: Evaluation of RANKL/OPG Levels in Gingival Crevicular Fluid at 1st and 3rd Months of Activation of NaOCl With Er,Cr YSSG Laser in Root Canal Treatment of Mandibular Molar Teeth With Periapical Lesions
Brief Title: Evaluation of RANKL/OPG Levels in Gingival Crevicular Fluid at 1st and 3rd Months of Activation of NaOCl With Er,Cr YSSG Laser in Root Canal Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Esin Özlek, Assoc.Prof, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10/15.12.2021
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Periapical Diseases
Keywords: Gingival cervicular fluidi; RANKL; OPG
MeSH Terms: conditions — Periapical Diseases

STUDY DESIGN:
Intervention Model Description: Group1: NaOCl, Er,Cr:YSSG will be activated by laser during the final irrigation; Group2 (control): Routine final irrigation procedure will be done, NaOCl will not be activated by any method) teeth will be divided into two main groups (n:15).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Er,Cr:YSSG laser (Active Comparator): NaOCl, Er,Cr:YSSG will be activated by laser during the final irrigation
  Interventions: Device: Er,Cr:YSSG laser; Device: Control
- Control (Active Comparator): Routine final irrigation procedure will be done, NaOCl will not be activated by any method.
  Interventions: Device: Er,Cr:YSSG laser; Device: Control

INTERVENTIONS:
Device: Er,Cr:YSSG laser — NaOCl, Er,Cr:YSSG will be activated by laser during the final irrigatio
Device: Control — Routine final irrigation procedure will be done, NaOCl will not be activated by any method)

SUMMARY:
Chronic Apical Periodontitis (CAP) is a disease caused by bacterial infection of the dental pulp and characterized by inflammation of the periradicular tissues. This disease is often the result of untreated caries and accompanied by the destruction of periapical bone and soft tissues, can cause tooth loss. Inflammatory periapical lesion is observed in the radiological examination of teeth diagnosed with Chronic Apical Periodontitis. This periapical lesion manifests as a host defense response to microbial challenge caused by infected pulp necrosis. Polymorphonuclear leukocytes, T and B lymphocytes, macrophages and plasma cells and many inflammatory cells are involved in host defense. These inflammatory cells, especially macrophages, mediate the immunological response seen in chronic apical periodontitis. Diagnosis and evaluation of apical periodontitis are made with conventional periapical radiographs. However, radiographic evaluation has some limitations. These limitations can be listed as the radiolucent area on the x-ray being related to the amount of bone loss caused by the lesion, the extent of the bone loss to the cortical bone, the variability of the bone structure in maxilla and mandibula, and the operator experience. The main goal in root canal treatment is to eliminate microorganisms and products in the root canal system with the irrigation agents which we use. NaOCl, which is frequently used for this purpose, is used alone or activated by Er,Cr YSSG laser. It has been reported that NaOCl, which is activated by laser, increases the elimination of microorganism in the root. The gingival crevicular fluid is an inflammatory exudate collected from the gingival sulcus. Peripheral body fluids, such as gingival crevicular fluid, can often be used as descriptors in acute and chronic inflammation. The collection of gingival crevicular fluid is a very simple and risk-free method for the patient. Biomarkers such as inflammatory mediators and neuropeptides can be detected in the gingival crevicular fluid of teeth with periodontal disease. At the molecular level, osteoclast activation is regulated by the triple molecule interaction of RANK, RANKL, and OPG. RANK (Receptor Activator of Nuclear Factor Kappa B) binds to its ligand, RANKL, while synthesizing both mature osteoclasts and its progenitor cells. RANKL provides osteoclast differentiation and activation. OPG (Osteoprotegerin) ligand is a decoy receptor for RANKL, thus inhibiting osteoclast differentiation.When the investigators look at the studies in the literature, there are many studies showing that the level of RANKL/OPG in the gingival crevicular fluid decreases with periodontal treatment. Also, when the investigators look at the studies on endodontic treatment, many mediators such as MMP-8, IL-8, Substance P, Neurokinin A and their changes after root canal treatment were examined. However, no study was found examining RANKL/OPG levels in gingival crevicular fluid after root canal treatment. At the same time, it is known that gingival crevicular fluid is used as a descriptive method in the determination of bone healing after periodontal treatment. However, in the literature, conventional radiological methods and tomography are seen as the most frequently used examination methods in the determination of bone healing after root canal treatment of lesioned teeth. The number of studies in which the gingival groove fluid collection method, which is much less invasive than these methods, is used as a descriptive method is quite limited. In line with this information, it is planned to conduct the research described below by examining the effect of activation with Er,Cr YSSG laser on the RANKL/OPG levels in the gingival crevicular fluid in the 1-3 month bone healing period after root canal treatment in lesioned teeth.

DETAILED DESCRIPTION:
The study is planned to be conducted on a total of 30 healthy patients, aged between 18-50 years, who were diagnosed and followed up in the Department of Endodontics, Faculty of Dentistry of Yüzüncü Yıl University. The sample size was calculated in the G*Power 3.1 program based on the data in the study of Arslan et al. In this study, the minimum required number of patients was determined as 30 by taking effect size 1.252193, alpha=0.05 and power=0.90. Mandibular first and second molars diagnosed with Chronic Apical Periodontitis will be included in the study group. Patients who do not have periapical lesions, have open apex, have a probing depth of more than 3 mm, and have bleeding during probing will not be included in the study group. RANKL and OPG levels in the gingival crevicular fluid will be determined using the ELISA test. RANKL and OPG levels in the gingival crevicular fluid of teeth with periapical lesions, which are indicated for root canal treatment, will be recorded with Periopaper (Oraflow, New York, NY).

Before taking a sample of gingival crevicular fluid, the tooth will be washed with water, dried and the plaque and deposits on it will be cleaned with cotton. Then, the tooth will be isolated with a cotton pellet and a suction, and a Periopaper (Oraflow, New York, NY) will be placed 1-2 mm into the gingival sulcus until slight resistance is felt, and a sample of gingival crevicular fluid will be taken after waiting for 30 seconds. Specimens contaminated with blood or saliva will not be included in the study. Then, these samples will be stored at -80°C. The access cavity will be opened to the teeth under local anesthesia with a 2 milliliter Ultracain D-S (Aventis, The Netherlands). The working length will be determined with a #15 K-files (Mani Inc, Tochigi, Japan) with the apex locator (DentsplyMaillefer, UK) and radiographic imaging.

The preperation of the root canals will be completed by ProTaperNext (DentsplyMaillefer, Baillagues, Switzerland) up to the X3 instrument as standard in each patient. 2 ml of 5.25% NaOCl solution will be used at each file change during preperation. During the irrigation process, a 2 milliliter dental injector and a 27 gauge dental needle tip will be used during preperation. The tip of the cannulas will be adjusted to be 1 mm shorter than the working length. Calcium hydroxide (Kalsin; Aktug Tic Bornova,Izmir, Turkey) paste is placed in the root canals after the preperation process and the tooth is temporarily closed with Cavit-G (3M ESPE, Seefeld, Germany). And the patient will be given an appointment 2 weeks later. When the patient comes to the second session appointment, the temporary restoration will be removed and the calcium hydroxide paste from root canals will be removed. Canals will be irrigated with 5 ml NaOCl 5.25% and 17% EDTA solution for the removal of calcium hydroxide. Then canals will reshaped with ProTaperNext X3 (DentsplyMaillefer, Baillagues, Switzerland). And then again 5 ml. NaOCl 5.25% and 17% EDTA solution will be used for irrigation to be ensured that calcium hydroxide is completely removed from the root canals. For final irrigation respectively 5 ml NaOCl %5,25 solution , 5 ml. % 17 EDTA solution and %5,25 NaOCl solution will be used. According to NaOCl activation (Group1: NaOCl, Er,Cr:YSSG will be activated by laser during the final irrigation; Group2 (control): Routine final irrigation procedure will be done, NaOCl will not be activated by any method) teeth will be divided into two main groups (n:15).

After final irrigation and activation procedure, root canals will be dried with sterile paper points, then all root canals will be obturated with sterile gutta-perchas and AH Plus root canal sealer (Dentsply DeTrey Gmbh, Konstanz, Germany) using the single-cone technique. Teeth with completed root canal filling will be restored with composite filling material to ensure coronal sealing. After the treatment, the patients in both groups will be called for control at periodically (1st month - 3rd month) and gingival crevicular fluid samples will be taken again with Periopaper (Oraflow, New York, NY). According to the results which is obtained with the ELISA test, the change in the RANKL and OPG levels in the gingival crevicular fluid of the patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons between the ages of 18 and 50 years
* Mandibular molar teeth that were diagnosed with periapical lesions

Exclusion Criteria:

* Pregnancy or lactation
* Patients who do not have periapical lesions,
* Teeth with immature/open apex
* A probing depth of more than 3 mm
* Bleeding during probing will not be included in the study group
* Teeth with root resorption

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
RANKL/OPG levels | 3 months
  RANKL/OPG levels in the gingival crevicular fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yıl University, Van, Turkey (Türkiye)

REFERENCES:
- [Background] Arslan H, Koseoglu S, Doganay Yildiz E, Arabaci T, Savran L, Yildiz DA, Veyisoglu G. Effect of intracanal diode laser application and low-level laser therapy on CGRP change. Braz Oral Res. 2019 Mar 18;32:e125. doi: 10.1590/1807-3107bor-2018.vol32.0125. PMID 30892373
- [Derived] Evrendilek F, Ozlek E, Meydan I. Effect of Er, Cr: YSGG laser-activated final irrigation on gingival crevicular fluid RANKL/OPG levels. Sci Rep. 2025 Dec 23. doi: 10.1038/s41598-025-33466-w. Online ahead of print. PMID 41436629